CLINICAL TRIAL: NCT01205984
Title: Efficacy and Tolerability of Systemic Methylprednisolone in Children and Adolescents With Chronic Rhinosinusitis
Brief Title: Systemic Methylprednisolone in Chronic Rhinosinusitis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ondokuz Mayıs University (Other)
Responsible Party: Fadıl Ozturk, Ondokuz Mayıs University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CRS-0655-IF
Record Dates: First submitted 2010-09-20; First posted 2010-09-21 (Estimated); Last update posted 2010-09-21 (Estimated); Status verified 2010-09

CONDITIONS: Chronic Rhinosinusitis; Children
Keywords: Chronic rhinosinusitis; Computed tomography scan; Methylprednisolone
MeSH Terms: interventions — Methylprednisolone; Tablets

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- oral methylprednisolone (Active Comparator)
  Interventions: Drug: methylprednisolone
- placebo (Placebo Comparator)
  Interventions: Drug: methylprednisolone

INTERVENTIONS:
Drug: methylprednisolone — Patients enrolled in the study were given either oral amoxicillin/clavulanate (AMX/C) or metylprednisolone (MP) (group MP) or AMX/C and placebo (group P) twice daily using a random allocation chart based on a table of random numbers. Oral AMX/C was administered 45/6.4 mg/kg/d (maximum 2000/285 mg/d) for 30 days for both groups. Oral MP was administered for the first 15 days: 1 mg/kg/d (maximum 40 mg/d) for 10 days, 0.75 mg/kg/d for 2 days, 0.5 mg/kg/d for 2 days, and 0.25 mg/kg/d for 1 day. Placebo tablets contained lactose and were of same size and color as MP tablets.
  Other Names: Prednol tablet; Augmentin suspension/tablet

SUMMARY:
The place of systemic corticosteroids in the treatment of children with chronic rhinosinusitis (CRS) remains unclear. We aimed to assess the effectiveness and tolerability of oral methylprednisolone (MP) as an anti-inflammatory adjunct in the treatment of CRS in children.Forty-eight children (age 6-17 years) with clinically and radiologically proven CRS were included. Patients were randomly assigned to either oral amoxicillin/clavulanate (AMX/C) and MP or AMX/C and placebo (P) twice daily for 30 days. Oral MP was administered for the first 15 days with a tapering schedule. Primary parameters were mean change in symptom and sinus computed tomography (CT) scan scores after treatment. Secondary study parameters were mean changes in individual symptom scores after treatment, relapse rate and tolerability. Forty-five patients completed the study, 22 received AMX/C and MP, and 23 AMX/C and P. Both groups demonstrated significant improvements in symptom and sinus CT scores, comparing baseline to end of the treatment (p<0.001). Methylprednisolone as an adjunct was significantly more effective than placebo in reducing CT scores (p=0.004), total rhinosinusitis symptoms (p=0.001) and individual symptoms of nasal obstruction (p=0.001), postnasal discharge (p=0.007), and cough (p=0.009). At the end of the treatment, 48% of the children in the P group still had abnormal findings in CT versus 14% in the MP group (p = 0.013). Therapy-related adverse events were not different between groups. Although insignificant, the incidence of clinical relapses was also less in the MP group (25%) compared to P group (43%) (p = 0.137). Oral MP is well tolerated and provides added benefit to treatment with antibiotics for children with CRS.

ELIGIBILITY:
Inclusion Criteria:All patients presented with nasal and/or postnasal purulence, and one or more of the following symptoms: nasal obstruction, cough, halitosis, headache, or facial pain/pressure. The diagnosis of CRS was made on the basis of sinonasal symptoms and signs present for a period of more than 3 months in the presence of abnormalities on coronal sinus CT scans.

-

Exclusion Criteria:Patients were excluded if they had used systemic corticosteroids in the last 2 months prior to the study, systemic antibiotics and inhaler or intranasal corticosteroids in the last 4 weeks prior to the study or if they had other respiratory disorders (cystic fibrosis, ciliary dyskinesia, nasal polyps, large adenoids, asthma), immune deficiency, systemic disease, gastro-esophageal reflux, aspirin sensitivity, and acquired or congenital sinonasal abnormalities, or a contraindication to corticosteroid use.

-

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 48 (Actual)
Dates: Start 2007-07; Primary Completion 2009-09 (Actual); Study Completion 2010-04 (Actual)

PRIMARY OUTCOMES:
Mean change in total symptom score and coronal CT score after treatment | One month
  Rhinosinusitis symptoms were assessed by the patients and their parents with the use of a visual analogue scale (VAS) rating symptoms from 0 (none) to 10 (most severe). A coronal sinus CT scanning was performed on all subjects before and at the end of the treatment. The scans were evaluated and scored according to the Lund-Mackay staging system.

SECONDARY OUTCOMES:
mean changes in individual symptom scores after treatment | One month
relapse rate | Six months
tolerability of oral methylprednisolone tablet | One month

CONTACTS AND LOCATIONS:
Overall Officials: Fadıl Ozturk, Principal Investigator — Ondokuz Mayıs University, Samsun, Turkey Gazi University,Ankara, Turkey; Ipek Turktas, Study Director — Gazi University, Ankara, Turkey
Locations (1):
- Gazi University Faculty of Medicine, Ankara, Turkey (Türkiye)